CLINICAL TRIAL: NCT02069769
Title: Ensuring Communication in Hospice by Oncology Study (ECHO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jennifer Temel, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-540
Record Dates: First submitted 2014-02-18; First posted 2014-02-24 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Ovarian Cancer; Cervical Cancer; Uterine Cancer; Head and Neck Cancer; Sarcoma; Melanoma
Keywords: Hospice Care; Head and Neck cancer; Gynecological Oncology; Sarcoma; Melanoma
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Cervical Neoplasms; Uterine Neoplasms; Head and Neck Neoplasms; Sarcoma; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- communication with oncology team (Experimental): oncology team will be prompted to contact family caregiver and/or patient twice weekly while the patient is receiving hospice care.
  Interventions: Behavioral: communication with oncology team

INTERVENTIONS:
Behavioral: communication with oncology team — Oncology team will contact patients and families via telephone at specific intervals

SUMMARY:
The goal of this study is to determine if scheduled communication with the oncology team through phone calls is helpful to caregivers with the transition to hospice care.

DETAILED DESCRIPTION:
There are four parts of the study. First, the participant will receive phone calls twice a week from the oncology team to check in with how the transition to hospice is going. Second, the participant may choose to have an appointment with the Massachusetts General Hospital oncology team to discuss any questions or concerns regarding cancer care or the transition to hospice. Third, each week of hospice care, the participant will be asked to complete a set of questionnaires at a time that is convenient for them either by phone or by email. These questions will ask the participant about their recent thoughts and feelings about their experience with hospice and as a caregiver. The questions will take less than 15 minutes to answer. Fourth, after hospice care has ended, the participant will be called by the oncology team to again check in and about a month later, the participant will also be contacted by phone to complete a set of questionnaires, again asking about their thoughts and feelings about your experience with hospice and as a caregiver.

For all of the questionnaires, the participant may skip any questions that the participant prefers not to answer. The responses will remain confidential and will be available only to study staff members who are trained in confidentiality and research ethics.

Additionally, during the research study, the investigators will obtain information from the participant's loved one's Massachusetts General Hospital electronic medical record that is relevant to the participation in the study for up to 6 months. If he/she has visited another hospital during this time, the investigator will also ask the participant for their permission to obtain the medical records from this visit.

The participant will not receive any compensation for this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patient Criteria

  -->18years of age) with a diagnosis of an incurable malignancy of the head and neck, gynecological oncology, sarcoma, or melanoma
  * Receiving oncology care at the MGH Cancer Center
  * Referral to home hospice services in previous five business days.
* Family Caregiver Eligibility Criteria:

  * Designated adult family/informal caregiver for an eligible patient who will provide the primary home care for the patient receiving hospice services
  * Ability to read and respond to questions in English or with the assistance of a translator
  * Access to telephone and/or computer to communicate with the oncology team and complete questionnaires
  * Willingness to complete weekly questionnaires via telephone or email.

Exclusion Criteria:

* Patient Exclusion Criteria:

  -- Referral to hospice services away from home (eg in nursing home or in an inpatient or residential setting)
* Family Caregiver Exclusion Criteria --Person is not the primary caregiver for the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the feasibility of implementing the Ensuring Communication in Hospice by Oncology Study (ECHO) intervention by patients' family caregivers and their oncology providers. | 2 Years
  ECHO will be considered feasible if greater than 70% of participants have > 50% of the scheduled phone contact with the oncology team during hospice care, which will be documented in the patient's medical record. Feasibility will also be demonstrated if greater than 70% of the family caregivers completing the questionnaires do so greater than 50% of the time they were scheduled. Finally, feasibility will also be demonstrated if caregivers are able to be contacted and decide upon participation within 5 days of patient hospice enrollment.

SECONDARY OUTCOMES:
Prospectively explore the satisfaction with the overall experience of family caregivers through questionnaires when receiving the ECHO intervention. | 2 Years
Prospectively explore rates of health service utilization in the patients receiving the ECHO intervention in terms of (1) hospice disenrollment; (2) hospitalization; and (3) emergency department visits | 2 Years
Prospectively explore the levels of stress of family caregivers through questionnaires when receiving the ECHO intervention. | 2 years
Prospectively explore decision making regret of family caregivers through questionnaires when receiving the ECHO intervention. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Temel, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States